CLINICAL TRIAL: NCT01434459
Title: Phase I Trial of Gemcitabine With TheraSphere® (Yttrium-90) in Patients With Hepatic Tumors of Pancreatobiliary Origin
Brief Title: Study of Gemcitabine With TheraSphere® (Yttrium-90)in Patients With Hepatic Tumors of Pancreatobiliary Origin
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: PI moved to different institution
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Bassel El-Rayes, Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00047233a; WCI1907-10 (Other: Other)
Record Dates: First submitted 2011-09-12; First posted 2011-09-15 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-05

CONDITIONS: Pancreatic Neoplasms; Cholangiocarcinoma
Keywords: Pancreatic neoplasms; Cholangiocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms; Cholangiocarcinoma | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gemcitabine with TheraSphere (Experimental)
  Interventions: Drug: Gemcitabine with TheraSphere

INTERVENTIONS:
Drug: Gemcitabine with TheraSphere — Gemcitabine dose will be escalated and combined with therasphere.
  Other Names: TheraSphere_radioembolization; Gemcitabine- Gemzar

SUMMARY:
Therasphere is a form of treatment that has been designed to selectively deliver radiation to the cancer within the patient's liver. This form of treatment has been used in a number of clinical trials and has been approved for use in the treatment of liver cancer.

The investigators want to test the safety of using Gemcitabine (a chemotherapy drug) with TheraSphere (radioactive beads that are injected directly into the blood vessel supplying the tumor in the liver) in patients with advanced pancreatobiliary tumors such as pancreatic cancer or cholangiocarcinoma (bile duct tumors) involving the liver.

DETAILED DESCRIPTION:
Patients with liver predominant cholangiocarcinoma or pancreatic cancer will be considered for the trial. The patients wre being treated in groups of thre patients. Each three patients receive a pre-specified dose of gemcitabine with full dose radioembolization using theraspheres. If no significant side effects are observed then three additional three patients will be treated with a higher dose of gemcitabine. The purpose to identify the highest dose of gemcitabine that can be safely combined with theraspheres.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic or cytologic diagnosis of pancreatic cancer or cholangiocarcinoma
2. Liver predominant disease defined as

   - Cholangiocarcinoma: liver disease should be unresectable

   - Limited extra hepatic metastasis defined as: i. Lung metastasis: 6 or less nodules with no nodule greater than 1.5 cm.

   ii. Abdominal lymph nodes iii. Pancreatic primary as long as the size is less than 4 cm in size iv. Bone metastasis
3. No prior systemic therapy for advanced stage disease
4. Measurable target tumors using standard imaging techniques
5. Lung shunting less than 20%
6. ECOG performance status 0-1 (See Appendix )
7. Age ≥ 18 years
8. No other investigational agents while on protocol
9. Signed informed consent

Exclusion Criteria:

1. Inadequate hepatic function: AST/ALT > five times upper limit of normal, Bilirubin >2.0 mg/dl or history of hepatic encephalopathy
2. Inadequate renal function Creatinine > 2.0 mg/dL
3. Inadequate bone marrow function: platelets < 100,000/mL or absolute neutrophil count <1500/mL
4. Contraindication to angiography
5. Prior external beam radiotherapy to the upper abdomen
6. Clinical evidence of peritoneal metastasis or ascites
7. Patients with extensive tumor replacement in the liver defined as >50% of liver involved with tumor
8. Any serious ongoing extra-hepatic disease such as infections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-09; Primary Completion 2014-01 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
The maximum tolerated dose of gemcitabine when given in combination with therasphere | 28 days
  Patients will receive full dose therasphere. The gemcitabine dose will start out low and the dose will increase after first 3 patients if no significant side effects are observed. The investigators will continue to increase the dose of gemcitabine as long as the investigators do not observe side effects or until we reach full dose of gemcitabine.

SECONDARY OUTCOMES:
Toxicities (side effects) experienced by patients on the trial | 90 days
  Any side effect experienced on the trial will be graded according to the grading system developed by the national cancer institute. The number of patients with each side effect will be calculated.
Tumor response rate when treated with gemcitabine and Therasphere using CT scan and F18-FDG-PET scan . | 78 days
  Patients will receive a PET CT prior to treatment and then another PET CT scan at completion day 78. Comparison of tumor size and uptake of FDG will be performed using standard RECIST criteria
The progression free of patients treated on the trial | 12 months
  The investigators will follow patients with serial cross sectional (CT or MRI) scans. If the tumor shows growth on the scan then the investigators will calculate the time it took for the tumor to grow.

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Kevin Kim, MD, Principal Investigator — Emory University Winship Cancer Institute; Bassel El-Rayes, MD, Principal Investigator — Emory University Winship Cancer Institute
Locations (1):
- Emory University, Atlanta, Georgia, United States